CLINICAL TRIAL: NCT06035003
Title: Mechanism of Mindfulness-Based Online Intervention in Enhancing Cognitive Flexibility: Thoughts as Thoughts
Brief Title: Mechanism of Mindfulness-Based Online Intervention in Enhancing Cognitive Flexibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230905
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iMIED+TAU group (Experimental): Internet-based Mindfulness Intervention for Emotional Distress (iMIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: Internet-based Mindfulness Intervention for Emotional Distress (iMIED)
- the TAU-only group (No Intervention): treatment as usual (TAU) group consisted of all medicinal and psychological treatments received between baseline and follow-up (about five months). Medicinal treatments included receiving Lorazepam, Olanzapine, Paroxetine Hydrochloride, Sertraline, etc. Psychological treatments included receiving cognitive behavior therapy or psychodynamic therapy.

INTERVENTIONS:
Behavioral: Internet-based Mindfulness Intervention for Emotional Distress (iMIED) — Internet-based Mindfulness Intervention for Emotional Distress (iMIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: iMIED+TAU group

SUMMARY:
Traditional offline interventions such as MBCT and MBSR have been implemented to treat patients with emotional disorders and obtained significantly improved clinical outcomes. However, these offline interventions require the involvement of a therapist expert in mindfulness and usually charge a high fee, which may not be accessible and cost-effective for lots of patients with psychological disorders. Fortunately, online self-help interventions can compensate for these disadvantages. Our research team has developed a self-help online mindfulness program targeting emotional distress (i.e., iMIED), which has been effective for individuals with emotional distress in a preliminary study. Since patients with emotional disorders usually suffer from emotional distress, the current study will apply this program to these patients, and investigate its auxiliary effects on patients' psychological and physical health.

The primary aim of the current study is to evaluate the effectiveness of iMIED for patients with emotional disorders. To do so, we will use a design in which patients who receive online mindfulness training (iMIED) except for treatment as usual (TAU) will be compared with patients who receive TAU alone. We expect the intervention to improve patients' psychopathological symptoms reported by the patients and the clinicians or the research team and increase their overall functioning, positive mental health, and physical health compared to TAU. In addition, previous studies have shown that mindfulness interventions improve psychological symptoms by improving cognitive flexibility. Therefore, the secondary aim of the study is to examine the mediating effect of cognitive flexibility on the relationships between mindfulness practice and improvements in outcome variables, and further explore the mechanism behind it.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet;
* Subjects with insufficient Chinese ability;
* Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire - Short Form during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Five Facet Mindfulness Questionnaire - Short Form is a self-reported questionnaire measuring mindfulness levels. Scores range from 20 to 100, with higher scores indicating higher levels of mindfulness.
Weekly changes of Patient Health Questionnaire during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Patient Health Questionnaire is a self-reported questionnaire measuring the degree of being troubled by various common physical symptoms. Scores range from 0 to 30.
  0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
Weekly changes of Chinese Perceived Stress Scale during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Athens Insomnia Scale during the intervention | [Time Frame: pre-intervention; weekly during the 7-week intervention; immediately post-intervention]
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.

SECONDARY OUTCOMES:
Change of Beck Anxiety Inventory | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Beck Anxiety Inventory is a self-reported questionnaire measuring anxiety. Scores range from 0 to 63, with higher scores indicating higher levels of anxiety.
Change of Beck Depression Inventory-II | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Beck Depression Inventory-II is a self-reported questionnaire measuring depression. Scores range from 0 to 63, with higher scores indicating higher levels of depression.
Change of Pittsburgh sleep quality Index | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Pittsburgh sleep quality Index is a self-reported questionnaire measuring sleep quality. Scores range from 0 to 21, with higher scores indicating lower levels of sleep quality.
Change of Insomnia Severity Index | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Insomnia Severity Index is a self-reported questionnaire measuring sleep quality. Scores range from 0 to 28, with higher scores indicating lower levels of sleep quality.
Change of Mindful Attention Awareness Scale | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Mindful Attention Awareness Scale is a self-reported questionnaire measuring mindfulness levels. Scores range from 15 to 90, with higher scores indicating higher levels of mindfulness.
Change of Quality of Relationship Index | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Quality of Relationship Index is a self-reported questionnaire measuring relationship quality. Scores range from 7 to 42, with higher scores indicating higher levels of relationship quality.
Change of Interpersonal Reactivity Index-C | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Interpersonal Reactivity Index-C is a self-reported questionnaire measuring interpersonal reactivity. Scores range from 0 to 88, with higher scores indicating higher levels of interpersonal reactivity.
Change of Intimacy Check and Evaluation Scale | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Intimacy Check and Evaluation Scale is a self-reported questionnaire measuring relationship intimacy. Scores range from 5 to 105, with higher scores indicating higher levels of relationship intimacy.
Moderation effect and possible changes of the Experience Questionnaire | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Experience Questionnaire is a self-reported questionnaire measuring decentering ability. Scores range from 20 to 100, with higher scores indicating higher levels of decentering ability.
Moderation effect and possible changes of the Emotion Regulation Questionnaire | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Experience Questionnaire is a self-reported questionnaire measuring emotion regulation ability. Scores range from 7 to 70, with higher scores indicating higher levels of emotion regulation ability.
Moderation effect and possible changes of the Cognitive Flexibility Inventory | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Cognitive Flexibility Inventory is a self-reported questionnaire measuring cognitive flexibility level. Scores range from 5 to 100, with higher scores indicating higher levels of cognitive flexibility.
Moderation effect and possible changes of the Thoughts as Thoughts Scale | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Thoughts as Thoughts Scale is a self-reported questionnaire measuring treating thoughts as thoughts ability. Scores range from 6 to 30, with higher scores indicating higher levels of treating thoughts as thoughts ability.
Moderation effect and possible changes of the Scale of Life Engagement | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Scale of Life Engagement is a self-reported questionnaire measuring life engagement. Scores range from 0 to 56, with higher scores indicating higher levels of life engagement.
Moderation effect and possible changes of the Self-Compassion Scale | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Self-Compassion Scale is a self-reported questionnaire measuring self- compassion. Scores range from 26 to 130, with higher scores indicating higher levels of self- compassion.
Moderation effect and possible changes of the Rumination- Reflection Questionnaire | [Time Frame: pre-intervention; 3 weeks into intervention; 5 weeks into intervention; immediately post-intervention]
  The Rumination- Reflection Questionnaire is a self-reported questionnaire measuring rumination- reflection level. Scores range from 5 to 60, with higher scores indicating higher levels of rumination- reflection.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Chen M, Hu A, Feng S, Hofmann SG, Liu X. Effect of cognitive flexibility in mindfulness intervention for emotional distress: Two randomized controlled trials. J Couns Psychol. 2025 Oct;72(5):581-597. doi: 10.1037/cou0000812. Epub 2025 Jul 14. PMID 40658552